CLINICAL TRIAL: NCT04301804
Title: A Phase I, Randomized, Single Center, Open-Label, Single Dose Pharmacokinetic Study of Reformulated SHR6390 Tablets Under Fasting Conditions in Healthy Caucasian Volunteers
Brief Title: A Trial of SHR6390 in Healthy Caucasian Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SHR6390-001AUS
Record Dates: First submitted 2020-03-01; First posted 2020-03-10 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2020-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: A total of 36 healthy volunteer subjects will be enrolled in this study. 12 subjects subjects will take a single dose of SHR6390 in each of the 3 dose cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose level 1 (Experimental): Subjects will be randomised to receive a single dose of SHR6390 at Dose level 1
  Interventions: Drug: SHR6390
- Dose level 2 (Experimental): Subjects will be randomised to receive a single dose of SHR6390 at Dose level 2
  Interventions: Drug: SHR6390
- Dose level 3 (Experimental): Subjects will be randomised to receive a single dose of SHR6390 at Dose level 3
  Interventions: Drug: SHR6390

INTERVENTIONS:
Drug: SHR6390 — a selective small-molecule CDK4/6 inhibitor

SUMMARY:
This is a Phase 1, single center, single dose, open-label clinical study to evaluate the pharmacokinetics, safety and tolerability of SHR6390 under fasting conditions in healthy caucasian volunteers

DETAILED DESCRIPTION:
The objective of this study is to determine the comparative pharmacokinetics, safety and tolerability of single oral dose of reformulated SHR6390 in healthy volunteers under fasting conditions.

Each subject will receive a single dose of SHR6390, blood samples will be collected before dosing and at various time points up to 144 hours after drug administration, safety and the statistical analysis of the pharmacokinetic data will be obtained from this study

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy Caucasian male and female subjects aged 18 to 45 years, inclusive at screening
* 2. Male body weight ≥50 kg, female body weight ≥45 kg, BMI between 19.0 and 29.0 kg/m2, inclusive
* 3. No clinically significant abnormalities in medical history, general physical examination, vital signs, laboratory tests
* 4. Female subjects agree not to be pregnant or lactating from beginning of the study screening and will maintain contraception for 90 days after trial completion
* 5. Males agree to use contraception with their female partner and refrain from donating sperm during the study and for at least 90 days after SHR6390 administration
* 6. Able and willing to abstain from caffeine- and xanthine-containing products, alcohol, grapefruit-related fruit juices, tobacco/nicotine-containing products, and alcohol for 48 hours prior to check-in until final PK blood sample
* 7. Able and willing to abstain from eating and drinking poppy seed-containing products and grapefruit-related fruits and juices
* 8. Able and willing to abstain from strenuous exercise
* 9. Willing and able to comply with all scheduled visits, study procedures, and provides written informed consent

Exclusion Criteria:

* 1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neuropsychiatric, or allergic disease
* 2. Had a severe infection, trauma or major surgery within 4 weeks of screening; plan to have a surgery during the trial
* 3. A past medical history of clinically significant cardiovascular conditions
* 4. Sitting systolic blood pressure (BP) ≥140 mmHg or <90 mmHg; diastolic BP ≥90 mmHg or <50 mmHg on a single measurement
* 5. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or any active systemic viral infection requiring therapy
* 6. Subject has a history of type 1 hypersensitivity to any medication
* 7. Evidence of substance abuse or a history of substance abuse in the last two years
* 8. Subject is positive for drugs of abuse,cotinine or alcohol at screening and check-in; may be repeated once at the discretion of the investigator
* 9. History of severe hypoglycemia
* 10. Subjects who use more than 5 tobacco or nicotine-containing products per day or will not abstain from using these products starting from at least 48 hours prior to check-in and during the study
* 11. History of regular alcohol consumption in the past 3 months exceeding an average weekly intake of 14 standard drinks
* 12. Use of medications affecting liver metabolism within 1 month prior to dosing
* 13. Treatment with an investigational drug within 3 months or 5 half-lives
* 14. Blood donation or loss of more than 200 mL of blood within 1 month of dosing or 400 mL of blood within 3 months, or 400 mL within 3 months.
* 15. Any other major illness/condition that, in the investigator's judgment, substantially increased the risk associated with the subject's participation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Number of subjects with laboratory tests findings of potential clinical importance | through study completion, an average of 1 year
Number of subjects with adverse events (AEs) | Screening up to study completion, an average of 1 year
Number of subjects with clinically significant abnormal ECG QT Interval | Screening up to study completion, an average of 1 year

SECONDARY OUTCOMES:
Pharmacokinetic - Cmax | 7 days
  Maximum observed plasma concentration (Cmax) of SHR6390
Pharmacokinetic - AUC∞ | 7 days
  Area under the concentration-time curve from time 0 to infinity of SHR6390
AUC from time 0 to the time of the last quantifiable concentration (AUClast) of SHR6390 | Day 1 pre-dose to Day 7 (144h) post-dose
Pharmacokinetic - AUClast | 7 days
  Area under the concentration-time curve from time 0 to time of last quantifiable concentration
Pharmacokinetic - Tmax | 7 days
  Time to Cmax of SHR6390
Pharmacokinetic - CL/F | 7 days
  Apparent clearance of SHR6390
Pharmacokinetic - Vz/F | 7 days
  Apparent volume of distribution during terminal phase of SHR6390
Pharmacokinetic - t1/2 | 7 days
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Melbourne, Western Australia, Australia